CLINICAL TRIAL: NCT06348563
Title: AGED Diagnostics Epigenetic Modifications of Liver Disease Assessment
Brief Title: AGED Diagnostics Liver Disease Assessment
Acronym: AGEDDX
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Active Genomes Expressed Diagnostics, Corp (Industry)
Collaborators: Arizona Clinical Trials (Unknown); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 7437787981
Record Dates: First submitted 2024-04-01; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: NASH With Fibrosis; NAFLD; Healthy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Health controls (Other): Diagnostic assessment
  Interventions: Diagnostic Test: AGED Multiple Target Assay in Healthy Controls
- NAFLD (Other): Diagnostic assessment. confirmation of diagnosis from liver biopsy is required.
  * NASH Diagnosis is on histological assessment from NASH CRN score:
    * NASH CRN score of ≤ 3 is classified as steatosis.
    * NASH CRN score of ≥ 5 is classified as NASH.
  * Participant samples can be subsequently diagnosed with CAP or MRI-PDFF to rule out NASH (or in rule in simple steatosis) but cannot be used to rule in NASH (as biopsy is required for confirmation).
  * All diagnostic criteria for participant at time of visit is requested.
  Interventions: Diagnostic Test: AGED Multiple Target Assay in NAFLD Participants
- Liver Fibrosis (Other): Diagnostic assessment, For fibrosis diagnosis and analysis, diagnostic tools can constitute zero or mild fibrosis (F0-F1), significant fibrosis (F2), and advanced fibrosis (F3-F4) in the presence or absence of NASH.
  * Participant samples can be diagnosed through non-invasive modalities such as but not limited to FIB4, ELF, PROC3, and/or imaging modalities such as but not limited to vibration controlled transient elastography (VCTE), magnetic resonance elastography (MRE), acoustic radiation force impulse (AFRI) or multiparameter imaging assessments.
  * All diagnostic criteria for participant at time of visit is requested.
  Interventions: Diagnostic Test: AGED Multiple Target Assay in Fibrosis Participants

INTERVENTIONS:
Diagnostic Test: AGED Multiple Target Assay in Healthy Controls — Analysis of blood based cfDNA/cfRNA biomarkers found at defined concentrations in participant samples that correlates to healthy controls
  Arms: Health controls
Diagnostic Test: AGED Multiple Target Assay in NAFLD Participants — Analysis of blood based cfDNA/cfRNA biomarkers found at defined concentrations in participant samples that correlates to NAFLD participants (defined as simple steatosis through NASH)
  Arms: NAFLD
Diagnostic Test: AGED Multiple Target Assay in Fibrosis Participants — Analysis of blood based cfDNA/cfRNA biomarkers found at defined concentrations in participant samples that correlates to liver fibrosis stage (F0-F4)
  Arms: Liver Fibrosis

SUMMARY:
Continue development of previously established methods to further validate candidate biomarkers that can discriminate steatosis from NASH and separately stage fibrosis from blood. The first assessment is to conduct test method verification to expand sample size to several hundred samples through whole genome sequencing methods. The second assessment is focused on biomarker validation by comparing targeted sequencing from patient plasma. Several sub- assessments will be conducted to support overall biomarker development efforts.

DETAILED DESCRIPTION:
Aim 1: Test Method Verification, Whole genome bisulfite sequencing assessment for liver tissue and plasma Conduct whole genome bisulfite sequencing in patient liver tissue and patient plasma to identified candidate biomarkers that can discriminate between steatosis and NASH, and separately conduct a comparative analysis of patient liver tissue and patient plasma samples to assess NASH encompassing NASH with mild fibrosis, NASH with significant fibrosis and NASH with advanced fibrosis. The purpose of each is to identify a set of markers that have biological relevance on the liver and then identify epigenetic biomarkers in plasma derived from liver tissue. Note: both a subset of NASH specific biomarkers and fibrosis specific biomarkers have been previously reported for technical feasibility.

Aim 2: Biomarker Validation, Targeted Epigenetic Sequencing Assessment Select top NASH specific biomarkers and top fibrosis specific biomarkers and design, develop and test probes to assess overall performance of each candidate biomarker in plasma. Conduct comparative analysis between various targeted sequencing and PCR based modalities. Candidate biomarker performance will be evaluated based on sensitivity, specificity, AUROC and reproducibility, among several other assessments.

ELIGIBILITY:
Inclusion Criteria:

* Participant with liver biopsy over the past 1-2 years are permissible for study inclusion.
* Participant is considered to be a "Healthy Subject" relative to any form of liver disease OR
* Participant is suspected of having one of the following diagnoses: metabolic syndrome, NAFLD, fibrosis/cirrhosis, cardiovascular disease, chronic kidney disease.

Exclusion Criteria:

* Participant is known to have HIV, Hepatitis B or Hepatitis C
* Participant has any other known form of chronic liver disease (aside from NAFLD/liver fibrosis)
* Participant has excess alcohol intake, excess alcohol is defined as participants that exceed an average 20g of alcohol daily for females (140g weekly intake) and average 30g of alcohol daily for males (210g weekly intake)
* Participant has had a bone marrow transplant at any time
* Participant is on anti-coagulation or anti-platelet therapy
* Participant is known to be pregnant
* Participant is unable to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Test Method Verification, Whole genome bisulfite sequencing assessment for liver tissue and plasma | 6-9 months
  Conduct whole genome bisulfite sequencing in patient liver tissue and patient plasma to identified candidate biomarkers that can discriminate between steatosis and NASH, and a separate assessment that can stage liver fibrosis.

SECONDARY OUTCOMES:
Biomarker Validation, Targeted Epigenetic Sequencing Assessment | 6-9 months
  Select top NASH specific biomarkers and top fibrosis specific biomarkers and design, develop and test probes to assess overall performance of each candidate biomarker in plasma through multiple targeted sequencing and PCR based modalities.

CONTACTS AND LOCATIONS:
Locations (1):
- AGED Diagnostics, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided